CLINICAL TRIAL: NCT02964156
Title: Effect of a Thin Customized Insole on Pain and Walking Ability in Rheumatoid Arthritis: A Randomised Study
Brief Title: Effect of a Thin Customized Insole in RA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Revmatismesykehuset AS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Revma nr 6
Record Dates: First submitted 2013-12-23; First posted 2016-11-16 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
Keywords: RA; Insole; Forefoot; Walking Ability; Pain
MeSH Terms: conditions — Arthritis, Rheumatoid; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Walking test using insoles (Experimental): Supersole
  Interventions: Other: Supersole
- Walking test not using insoles (Experimental): no intervention
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Supersole — A 4-mm thin, individually customized insole of a malleable plastic material (CI-Core®) with synthetic textile material on the upper side.
  Arms: Walking test using insoles
Other: No intervention — No intervention
  Arms: Walking test not using insoles

SUMMARY:
50-90% of patients with RA reports foot problems and the metatarsophalangeal joints of the forefoot are most frequently afflicted. Studies shows that foot problems can influence negatively on the walking function, physical activity and quality of life. Different foot orthoses and insoles are used as an intervention. Studies find that different insoles do have effect on pain, but there are no or minor effect on walking ability. The literature reports a further need for research and indicates the importance of studies on the effects of cost-effective insoles for patients with RA.

Custom-built insoles takes time and are often expensive, and many patients, especially women, do not wear them since they often do not fit the shoes they prefer to wear. In this study, a 4-mm thin, flat insole of a malleable plastic material (CI-Core®) with synthetic textile material on the upper side is customized to provide support for the transverse and longitudinal arches of the foot to reduce pressure on painful joints. The insole is easily customized and ready for use the same day. The purpose of this study was to determine whether this insole can reduce foot pain and increase walking distance in patients with RA and forefoot pain.

An experimental study was performed on patients with RA and forefoot pain in either one or both feet. The patients walked as fast as they could in 6 minutes (6MWT) with either insoles (situation A) and without insoles (situation B). The order of situation A and B was randomized, and the assessor was blinded for the order of the two situations. Both tests were conducted the same day. After each test round, the patient was asked to register pain in the foot and perceived exertion. A telephone interview was conducted one year after the effect study to examine whether the insoles were still being used.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis Rheumatoid Arthritis
* Foot pain while walking
* Positive Gaenslens sign in forefoot
* Native Norwegian speaking

Exclusion Criteria:

* Cognitive dysfunction
* Problems reading
* Problems in walking due to problems han the foot such as in ankel, knee or hip

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Pain intensity measured using Visual Analog Scale (VAS) | Change between test situation A and B (or B and A). A: Walking test using insoles. B. Walking test not using insoles. There is a 20 minute break between the two situations.
  Pain is measured using Visual Analog Scale (VAS)
Walking ability measured using the 6-minute walking test | Change between test situation A and B (or B and A). A: Walking test using insoles. B. Walking test not using insoles. There is a 20 minute break between the two situations.
  Walking ability is measured using the 6-minute walking test

SECONDARY OUTCOMES:
perceived exertion measured using Borg CR10 scale | Change between test situation A and B (or B and A). A: Walking test using insoles. B. Walking test not using insoles. There is a 20 minute break between the two situations.
  Perceived exertion is measured using Borg category ratio scale (Borg CR10)

CONTACTS AND LOCATIONS:
Overall Officials: Knut Mikkelsen, MD, Study Chair — Revmatismesykehuset AS, Lillehammer, Norway

IPD SHARING:
Plan to Share IPD: No